CLINICAL TRIAL: NCT01944436
Title: Lewy Body Spectrum Disorders: Investigating Neuropsychiatric Benefit and Adverse Effects in Response to Cholinesterase Inhibitors Using Genetics and Brain SPECT
Brief Title: A Genetic and Perfusion Study of Response to Cognitive Enhancers in Lewy Body Disease
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Mario Masellis, Clinician-Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: LBD-312-2006
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Lewy Body Disease
Keywords: Pharmacogenomics; Dementia with Lewy bodies; Adverse events; Polymorphisms; Acetylcholinesterase; Parkinson's Disease Dementia; Cognitive enhancers; Clinical efficacy; Cytochrome P450; Butyrylcholinesterase
MeSH Terms: conditions — Lewy Body Disease; Pain; Butyrylcholinesterase deficiency | interventions — Cholinesterase Inhibitors; Rivastigmine; Donepezil; Galantamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Functional and tag SNPs in the following genes will be assessed:
  acetylcholinesterase (ACHE); butyrylcholinesterase (BCHE); M1 muscarinic receptor (CHRM1); alpha7-nicotinic receptor (CHRNA7); Apolipoprotein E (ApoE); Cytochrome P450 2D6 (protein: CYP2D6 /gene: CYP2D6); CYP3A4; all genes related to blood pressure disregulation, white matter changes found on neuroimaging, and genes related to Lewy Body Spectrum disorders in general.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease Dementia: Participants in the Parkinson's Disease Dementia group:
  * Must be taking a stable parkinsonian medication
  * Must have a diagnosis of clinically definite Parkinson's disease >1 year prior to cognitive deficit with at least two of the following symptoms: asymmetric resting tremor, rigidity or bradykinesia, and definite motor response to dopaminergic agents.
  * Response to cholinesterase inhibitor over a period of six months will be monitored.
  Interventions: Drug: Cholinesterase Inhibitors (Rivastigmine, Aricept, Galantamine)
- Dementia with Lewy Bodies: Participants in the Dementia with Lewy Bodies group:
  * Diagnosis of clinically probable or possible Dementia with Lewy bodies with at least 1 of the following: Marked fluctuations in cognition, visual hallucinations or spontaneous parkinsonism.
  * Response to cholinesterase inhibitor over a period of six months will be monitored.
  Interventions: Drug: Cholinesterase Inhibitors (Rivastigmine, Aricept, Galantamine)

INTERVENTIONS:
Drug: Cholinesterase Inhibitors (Rivastigmine, Aricept, Galantamine)

SUMMARY:
Lewy body spectrum disorders are a common group of neurodegenerative diseases that cause memory loss, behavioural and motor disabilities that impair quality of life. Cognitive enhancers help people afflicted with these conditions. However, some people do not benefit from this treatment, while others experience serious side effects. Side effects and poor response lead to hospitalization and early institutionalization. Pharmacogenomics, the study of how DNA variation can influence drug effects, will be combined with functional changes in brain imaging in response to cognitive enhancers in patients with Lewy body disease. The goal is to develop a predictive test that can be administered in the clinic to aid physicians' choice of initial medication. This can reduce health care costs and improve treatment to Canadians suffering from these devastating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients with a Lewy body spectrum disorder includes: age > 50 years; and mild-moderate dementia (Mini-Mental State Exam [MMSE] > 9); contact on at least four of seven days/week with a responsible caregiver; Hoehn & Yahr stage ≤ 4.

Exclusion Criteria:

* age < 50; Severe dementia (MMSE < 9); contact < 4 days a week with a responsible caregiver; Hoehn & Yahr stage > 4.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2006-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in perfusion brain SPECT at 6 months | 0 and 6 months
Change from baseline in neuropsychological assessment scores at 6 months | 0 and 6 months

SECONDARY OUTCOMES:
Volumetric Brain MRI | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada